CLINICAL TRIAL: NCT01000467
Title: A Randomized, Open-label, Single-center Clinical Trial to Evaluate the Safety and Pharmacokinetics of Probucol by Multiple Administration in Healthy Male Subjects
Brief Title: Pharmacokinetics Study for Probucol
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Korea Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 009-KOB-0801i
Record Dates: First submitted 2009-10-18; First posted 2009-10-23 (Estimated); Last update posted 2022-03-04 (Actual); Status verified 2009-10

CONDITIONS: Healthy
Keywords: PK assessment for healthy male volunteer; Healthy male subjects aged 20 to 40 years
MeSH Terms: interventions — Probucol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 2 (Active Comparator): Group 2(probucol 500mg BID)
  Interventions: Drug: probucol
- 1 (Active Comparator): Group 1(Probucol 250mg)
  Interventions: Drug: probucol
- 3 (Active Comparator): Group 3(Probucol 500mg once daily)
  Interventions: Drug: probucol

INTERVENTIONS:
Drug: probucol — group 3: 250 mg 1 tablet in the morning and evening
  Other Names: Brand name: Lorelco
  Arms: 3
Drug: probucol — group 1: 250 mg
  Other Names: lorelco
  Arms: 1
Drug: probucol — group 2: 250 mg 2 tablets at once in the morning
  Other Names: Lorelco
  Arms: 2

SUMMARY:
To evaluate the safety and pharmacokinetics of probucol by multiple oral administration in healthy male subjects.

DETAILED DESCRIPTION:
To evaluate the safety and pharmacokinetics of probucol by multiple oral administration of one 250-mg probucol tablet once daily after breakfast (250 mg/day), two 250-mg probucol tablets once daily after breakfast (500 mg/day), and one 250-mg probucol tablet twice daily after breakfast and dinner (500 mg/day) for 14 days in healthy male subjects.

ELIGIBILITY:
Inclusion criteria

* Korean
* Male
* Age from 20 to 40 years at time of informed consent
* BMI more than 19.0 and less than 25.0
* Subjects who meet the following criteria at the time of the screening
* Subjects with ECG results without AV block and with both of qTc and QRS width within the standard values

Exclusion criteria

* History or clinical evidence of significant medical history
* Present or previous significant drug allergy to any prescription or OTC medication

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2009-02; Primary Completion 2009-08 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Plasma pharmacokinetic (PK) parameters: Auc, Cmax etc. | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-Sang Yoo, MD, PhD, Principal Investigator — Clinical Trial Center, Seoul National University Hospital
Locations (1):
- Seoul national univeristy, Seoul, South Korea